CLINICAL TRIAL: NCT05667311
Title: Evaluation of Autonomic Function Deficits in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Autonomic Function in Patients With COPD
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Guy Joos, Prof. Eric Derom, University Hospital, Ghent
Other Study IDs: B670201628572
Record Dates: First submitted 2016-08-16; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Autonomic Function in Patients With Chronic Obstructive Pulmonary Disease
Keywords: Genetics; COPD; Autonomic nervous system
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ECG — Finapres electrocardiography machine

SUMMARY:
Conduct an in-depth evaluation of autonomic function using a validated tests, assess genetic aspects of autonomic failure, and determine the correlation between of autonomic function failure and other clinical variables in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a highly prevalent systemic disease that is caused by both environmental determinants and genetic risk factors. Patients with COPD also present with several comorbidities affecting their overall health status (Berndt et al, 2012). The investigators have demonstrated from recently conducted systematic reviews that patients with COPD have significant impairments in autonomic function (Mohammed et al, 2015). Our ongoing hospital survey (preliminary results) also indicates these patients have significant autonomic complaints (symptoms). Consequently, the objectives of this present study are to; i) conduct an in-depth evaluation of autonomic function using a validated battery of tests, (ii) assess genetic aspects of autonomic failure, and (iii) to determine the correlation between of autonomic function failure and other clinical variables in patients with COPD.

Based on the experience of our group (PhD- De Wandele, 2014), the investigators will evaluate the cardiovascular function (reflexes) in patients with COPD of different GOLD stages. The recruitment will be based on our recent questionnaire study. The patients will be evaluated by four validated tests. The first test is the HRV at rest. In this test, the ECG during 30 minutes will be registered while the patient lies supine. The R-R intervals analysis will be evaluated by time (mean and standard deviation (SD) and other derived parameters such as SDNN) and frequency (Fast Fourier analysis to measure high frequency, low frequency bands and the ratio of HF/LF) domain parameters. The second test is the deep breathing maneuver. This test will be based on the phenomenon of respiratory arrhythmia. Here, patients will be asked to breath in and out at an imposed rhythm (8 cycles of 5 seconds in and 5 seconds out) that will be displayed on a screen (laptop). For this test, changes of heart rate (ECG) at breathing in and breathing out will be analyzed to ascertain its impact on parasympathetic activity. The third test is the valsalva manoeuver (which is evoked by blowing into a tube at a pressure between 40 and 50 mmHg for 15 seconds/3 trials). During this test (ECG recordings), the valsalva ratio (parasympathetic measure) and the 4 phases of blood pressure response (sympathetic reactivity) will be calculated and quantified (Novak, 2011). The adrenergic, vagal and global baroreflex sensitivity parameters will also be calculated (Schrezenmaier et al. 2007) from the ECG recordings. The fourth and last test is the head up tilt test. Here, the patient after 5 minutes of rest in supine position will be tilted rapidly to 60°. Due to redistribution of the blood in the body, this test is normally expected to evoke changes in blood pressure and heart rate that will be compared with the baseline measures. The tilt test (position) will last about 20 minutes. The initial orthostatic (hypotension) status will be taken into account.

In the end, the investigators will calculate a "composite autonomic severity score" (CASS) based on cardiogenic and adrenegic functions thats will be derived from tests. the CASS results will range from 0 (no autonomic deficit) to 10 (maximal deficit). Also, the CASS score will be associated with different parameters. These include anthropometric measures (BMI, weight, height, fat free mass and fat mass), disease phenotyping (lung function (tiffeneau-index, breathing frequency, ventilatory effort, dyspnea, number of exacerbations, disease progression, anxiety and subjective well-being) and medication usage.

This study also has a genetic aspect that will be carried out concurrently. Here, the investigators aim to determine the prevalence of autonomic failure genes in these patients and also correlate same with autonomic performance. For this, venous blood samples will be collected by a a nurse. These samples will be relayed to the medical genetics Department for DNA extraction and evaluation (polymorphisms). The evaluation will be based upon identification of autonomic failure genes that were earlier reported by Mathias & Bannister ( 2013). These genes include α2b-adrenergic receptor (5ADRA2B), dopamine receptor D4, Solute carrier family 6 (neurotransmitter transporter noradrenaline)-member 2, ........ This part of the study will be done in collaboration with the Medical Genetics Centre of the University Hospital Ghent.

In total, the investigators are aiming to recruit 50 patients.

ELIGIBILITY:
Inclusion Criteria:

Stable COPD Ambulant

Exclusion Criteria:

* Recent hospitilization (3 months) Recent exacerbation (3 months) Other chronic systemic diseases (eg CHF, DM)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD attending the respiratory medicine department or the pulmonary rehabilitation division of Ghent University Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses orthostatic intolerance
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses autonomic symptoms
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses secretomotor symptoms
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses gastrointestinal symptoms
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses urinary symptoms
Autonomic symptom score (COMPASS 31) questionnaire | 1 hour
  Asses pupillomotor symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided